CLINICAL TRIAL: NCT04400240
Title: Care Coordination Approaches to Learning Lupus Self-management
Acronym: CALLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Edith Williams, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00070647
Record Dates: First submitted 2020-05-08; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): complete questionnaires and phone sessions
  Interventions: Behavioral: CALLS
- Control (No Intervention): complete questionnaires only

INTERVENTIONS:
Behavioral: CALLS — The CALLS program will consist of 12 weeks of service delivery that will include one standard educational session by telephone or in-person meeting every week. The weekly educational session will be generally structured in three parts: introduction, structured education, and problem solving. Weekly content will be adapted from the twelve modules of the Peer Approaches to Lupus Self-management (PALS) study, and further tailored according to prominent barriers to care in the scientific literature. Content will include: 1) Medication adherence; 2) Communication with provider; 3) Patient engagement; 4) Recognizing and treating depression; 5) Overcoming socioeconomic barriers; 6) Social Support network; 7) Appointment/ Lab adherence; and 8) Transportation.
  Arms: Intervention

SUMMARY:
The Care-coordination Approach to Learning Lupus Self-Management (CALLS) study was designed to examine whether modeling and reinforcement from a lay patient navigator/care coordinator improves disease self-management, indicators of disease activity, health related quality of life (HRQOL), and 30-day readmission in SLE inpatient admissions. We recruited 30 patients (~15 questionnaires and phone sessions and 15 questionnaires only) with active SLE upon hospital admittance at the Medical University of South Carolina (MUSC). The lay patient navigator/care coordinator was trained to deliver intervention content by twelve weekly telephone sessions carried out across the course of the study. All participants were assessed using validated measures of patient reported outcomes at baseline, mid-intervention (6 weeks post-enrollment), and immediately following the intervention (12 weeks post-enrollment). Outcomes for patients who agreed to phone sessions were compared with the outcomes of patients who opted to participate in questionnaires only. The study lasted 12 months, with recruitment and enrollment over 6 months, 3 months for intervention delivery and 3 months for data analysis.

DETAILED DESCRIPTION:
Overview of Study Design. The Care-coordination Approach to Learning Lupus Self-Management (CALLS) study is a double arm, pre-post pilot designed to examine whether modeling and reinforcement from a lay patient navigator/care coordinator improves disease self-management, indicators of disease activity, health related quality of life (HRQOL), and 30-day readmission in SLE inpatient admissions. We will recruit 40 patients (20 questionnaires and phone sessions and 20 questionnaires only) with active SLE upon hospital admittance at the Medical University of South Carolina (MUSC). The lay patient navigator/care coordinator will be trained to deliver intervention content by twelve weekly telephone sessions carried out across the course of the study. All participants will be assessed using validated measures of patient reported outcomes at baseline, mid-intervention (6 weeks post-enrollment), and immediately following the intervention (12 weeks post-enrollment). Outcomes for patients who agree to phone sessions will be compared with the outcomes of patients who opt to participate in questionnaires only. The study will last 12 months with recruitment and enrollment over 6 months, 3 months for intervention delivery and 3 months for data analysis.

Study Population. The target population for this study will be SLE inpatient admissions at MUSC. There are approximately 35 SLE and Scleroderma hospital admissions each month, so it is expected that over a 3-month recruitment period, we will be able to recruit 40 participants (20 questionnaires and phone sessions and 20 questionnaires only).

Recruitment of Lay Patient Navigator/Care Coordinator The PI will identify a suitable lay patient navigator/care coordinator based on their maturity, emotional stability, and verbal communication skills. Suitable candidates will have at least a high school diploma or equivalency with at least one year of patient care experience in a health care facility; or a Certified Nursing Assistant; or successful completion of a Nursing Assistant or Medical Assistant course at an accredited institution or equivalent training; or EMT or Paramedic certification; or a Bachelor's degree. They will possess the ability to understand and implement a variety of detailed instructions in the execution of therapeutic procedures and the ability to make accurate physical observation of patients.

Recruitment of SLE patients Admitted SLE patients will be referred by their physician for participation in the study, who will provide a letter that will explain the study and provide participants a number to call if they have questions or concerns prior to agreeing to participate. Participants who indicate interest in the study will be immediately screened for eligibility, and if eligibility criteria are met, informed consent will be obtained. Once a patient has been consented, they will be randomized to membership in one of the two study arms. assigned to the intervention (complete questionnaires and phone sessions) or control (complete questionnaires only) arm, and the rest of the recruitment visit will include baseline self-report assessments and scheduling of phone sessions (if applicable).

Phone sessions: The CALLS program will focus on enhancing the health of SLE patients, with emphasis on patient empowerment and promoting proactive participation in health care. Recruitment and enrollment will occur on a rolling basis, and the program will consist of 12 weeks of service delivery that will include one standard educational session by telephone or in-person meeting every week. The weekly educational session will be generally structured in three parts: introduction, structured education, and problem solving. Weekly content will be adapted from the twelve modules of the Peer Approaches to Lupus Self-management (PALS) study, and further tailored according to prominent barriers to care in the scientific literature. Content will include: 1) Medication adherence; 2) Communication with provider; 3) Patient engagement; 4) Recognizing and treating depression; 5) Overcoming socioeconomic barriers; 6) Social Support network; 7) Appointment/ Lab adherence; and 8) Transportation. The lay patient navigator/care coordinator will respond to individual patient needs by tailoring intervention content to personal requirements and facilitating care coordination and will be able to address insurance, financial, and logistical issues (e.g., transportation, appointment scheduling, child or elder care), while providing understandable health education that may lessen fears of SLE diagnosis and treatment. Lay patient navigator/care coordinator activities will be guided by frequent self-report assessments, which will help to identify patient concerns across multiple domains, triage patients to appropriate resources, and ultimately overcome barriers to health care. The lay patient navigator/care coordinator can use baseline data collected prior to phone sessions to describe preliminary patient themes (i.e., disease activity and damage, depression, medication adherence, communication with provider, patient engagement) and subsequent assessments can be used to track progress.

Data Collection Schedule. Study questionnaires were carefully chosen based on available evidence of previous validation and their ability to measure key elements of the study aims. The primary method of data collection will be face-to-face interview. All study visits will take place in an MUSC affiliated hospital, the Research Nexus or comparable private location on the campus of MUSC. Indicators of medication adherence will be extracted from the electronic medical records. Financial data will be extracted from the research data warehouse for historical and patient-specific data for cost effectiveness. The MUSC REDCap system will be used for data management.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission for SLE-related issue;
2. clinical diagnosis of systemic lupus erythematosus (SLE) from a physician;
3. 18 years of age or older;
4. able to provide informed consent and take part in ongoing assessment/evaluation activities (self-reported questionnaires);
5. able to commit to duration of study (3 months);
6. able to communicate in English; and
7. have an active phone line (landline or cell phone) for the duration of the study, if agreeing to phone sessions with the lay patient navigator/care coordinator.

Exclusion Criteria:

1. cognitive impairment;
2. acute decompensation of chronic conditions precluding participation;
3. conditions that preclude participation in assessments (e.g. blindness or deafness); and
4. terminal illness or life expectancy less than 6 months as evaluated by physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Self-management measured using the Patient Activation Measure (PAM) | Baseline to post-intervention, at 12 weeks
  The Patient Activation Measure (PAM) assesses an individual's knowledge, skill, and confidence for managing their health and healthcare. Individuals who measure high on this assessment typically understand the importance of taking a proactive role in managing their health and have the skills and confidence to do so. The PAM survey measures patients on a 0-100 scale and can segment patients into one of four activation levels along an empirically derived continuum, including "Believes Active Role Important", "Confidence and Knowledge to Take Action", "Taking Action", and "Staying Course Under Stress". Each activation level reveals insight into an array of health-related characteristics, including attitudes, motivators, behaviors, and outcomes.
Satisfaction in Quality of Life as assessed by the LUP-QOL (Lupus Quality of Life Questionnaire) | Baseline to post-intervention, at 12 weeks
  Quality of life will be assessed by using The LUP-QOL (Lupus Quality of Life Questionnaire), which assesses areas of the participant's life that may be affected by lupus. The score ranges from 0-100. A score of '0' indicates the lowest quality of life, and a score of 100 indicates the best quality of life.

SECONDARY OUTCOMES:
30-day readmission | Baseline to post-intervention, at 12 weeks
  Change in cost due to readmission. Costs will include total charges associated with any healthcare encounters at the Medical University of South Carolina.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Results presented in peer-reviewed publications

REFERENCES:
- [Derived] White AA, Ba A, Faith TD, Ramakrishnan V, Dismuke-Greer CL, Oates JC, Williams EM. The Care-coordination Approach to Learning Lupus Self-Management: a patient navigator intervention for systemic lupus inpatients. Lupus Sci Med. 2021 May;8(1):e000482. doi: 10.1136/lupus-2021-000482. PMID 33975925